CLINICAL TRIAL: NCT06500338
Title: Determining the Dose Response Profile of the Headward Fluid Shift During Varying Gravity Levels
Acronym: AG2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Aeronautics and Space Administration (NASA) (U.S. Federal Agency)
Collaborators: NOVESPACE (Merignac, France) (Unknown); European Space Agency (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00000508
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Healthy
MeSH Terms: interventions — Weightlessness

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Preflight Seated (No Intervention): Preflight control at 1 Gravity level (G), seated. Data collection of Internal Jugular Vein (IJV) area, IJV pressure, and Doppler blood flow.
- Preflight Supine (No Intervention): Preflight control at 1 Gravity level (G), supine. Data collection of Internal Jugular Vein (IJV) area, IJV pressure, and Doppler blood flow.
- inflight reduced gravity measures (Experimental): inflight experimental at 0 Gravity levels (G), 0.25G, 0.5G, and 0.75G. Data collection of Internal Jugular Vein (IJV) area, IJV pressure, and Doppler blood flow.
  Interventions: Procedure: free-fall

INTERVENTIONS:
Procedure: free-fall — The aircraft will fly in parabolas that initially produce increased gravity (1.8-G, "hypergravity"), followed by ~20-50 second periods of partial gravity or weightlessness. Flights which produce partial gravity (0.25-, 0.50-, and 0.75-gravity) generally will consist of 31 parabolas (at least 10 parabolas at each gravity level), and flights that produce weightlessness generally will consist of 16 parabolas.
  Other Names: parabolic flight; partial gravity; weightlessness
  Arms: inflight reduced gravity measures

SUMMARY:
Parabolic flight provides a unique opportunity to evaluate the acute changes associated with varying levels of gravity and to describe how key venous parameters change at levels less than normal Earth gravity. Characterizing these changes in response to varying G-levels is an important step in determining what G-level may be required to reverse weightlessness-induced fluid shifts and thus serve as a viable countermeasure during long-duration spaceflight. Further, these results will inform National Aeronautics and Space Administration (NASA) whether there might be a lower risk of Spaceflight Associated Neuro-ocular Syndrome (SANS) and Venous Thromboembolism (VTE) during extended stays on the Moon and Mars.

DETAILED DESCRIPTION:
Subjects first will be studied for baseline data collection (BDC) on Earth in a 1 gravity-level (G) environment while seated and supine. During baseline data collection, the operator will identify the proper location of the internal jugular vein measurement (below the confluence of the internal jugular vein and superior thyroid vein) using ultrasound and mark this location with a marker so subsequent scans can be taken in the same location. Thereafter, six electrocardiogram electrodes will be adhered to the skin of the chest and connected to the ultrasound machine and to a data recording system. A small blood pressure cuff will be placed around one finger; blood pressure also will be recorded continuously. The blood pressure cuff will be inflated preflight during baseline data collection and inflight during the parabolas. Baseline ultrasound images of the internal jugular vein will be acquired in the seated and supine positions on the ground. Measurements will include 2D ultrasound of the right and left internal jugular veins for measurement of cross-sectional area and pressure, and Doppler ultrasound of the right and left internal jugular veins for flow characterization.

Anti-motion sickness medication is distributed to flying participants at their discretion. Participants board the Airbus A310 aircraft fasten seatbelts for takeoff. After takeoff, the pilots fly the aircraft to a specific air zone where the parabolas will take place. With other members of the participant's group, participants will then move to the area of the cabin in which data will be collected. Participants will receive instructions from Novespace to maintain safety during the parabolic flight.

The aircraft will fly in parabolas that initially produce increased gravity (1.8-G, "hypergravity"), followed by ~20-50 second periods of partial gravity or weightlessness. After that, there will be another pull-up (hypergravity) to complete the parabola. The plane then will fly in normal horizontal flight for a few minutes before repeating the parabolic flight path again. The pilots will perform this sequence of maneuvers many times. The number of times, the level of reduced gravity, and the order of reduced gravity exposures will depend upon the flight plan for that day. Subjects will be informed of the flight plan in the pre-mission briefing conducted by Novespace. Flights which produce partial gravity (0.25-, 0.50-, and 0.75-gravity) generally will consist of 31 parabolas (at least 10 parabolas at each gravity level), and flights that produce weightlessness generally will consist of 16 parabolas. The total flight time from take-off to landing is approximately 2-3 hours.

During the flight, subjects will be seated in a specially designed chair with a seatbelt, and the ultrasound operator will be seated to the right and front of them facing the subject. Measurements will be taken multiple times during partial gravity or weightlessness and during level flight. Subjects are requested to minimize movements during the ultrasound measurements so that accurate measurements can be obtained. Also, subjects will be encouraged to minimize any movements during periods of increased gravity ("pull-out", "pull-up") in order to prevent motion sickness.

After the data collection is completed, subjects will be disconnected from the hardware, and electrodes can be removed. While subjects may experience fatigue, tiredness, and motion sickness from participating in parabolic flight, there will be no direct effects from the ultrasound measurements, except for perhaps skin irritation from the electrodes.

During the consent process prior to collection of video or still images, we will ask for consent as designated on the Research Consent Form. Novespace will photograph or film participants in Novespace facilities, including the aircraft, and use those images for the purposes of promotion and communication. Also, photos or video recordings of test subjects may be collected by the investigator team during the experiment. These photos may be used in future presentations or publications to demonstrate procedures used during the flight study.

ELIGIBILITY:
Inclusion Criteria:

* In coordination with the parabolic flight company, Novespace, healthy volunteers from the population that are 25-55 years old without a history cardiovascular disease will be recruited for this study. In order to participate, subjects must be able to follow instructions in English.
* Participants must be age 18 years or older, hold a French or European Health Insurance Card, and provide medical certification of fitness for flight to NOVESPACE (i.e., NOVESPACE Parabolic Flight Medical Aptitude Certificate) completed by their medical doctor or an Authorized Medical Examiner.
* Participants must meet medical criteria and provide certification of fitness for flight to NOVESPACE (i.e. NOVESPACE Parabolic Flight Medical Aptitude Certificate) completed by their medical doctor or an Authorized Medical Examiner.

Exclusion Criteria:

* NOVESPACE exclusion criteria includes:
* Those with certain heart and lung conditions
* dizziness
* certain inner ear conditions
* severe motor disability or impaired bone density
* psychosis
* mental disability prohibiting emergency evacuation
* epilepsy
* certain neurological diseases
* fear of heights/flying
* debilitating anxiety and panic attacks
* claustrophobia, women who are pregnant
* certain gastrointestinal conditions
* those taking certain medications are ineligible to participate
* An individual's overall medical fitness for flight is assessed and certified by a medical doctor or Authorized Medical Examiner.
* Pregnant women are not eligible to participate in this study.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2024-04-17 (Actual)

PRIMARY OUTCOMES:
Bilateral Internal jugular vein blood flow characterization | 2-3 hours
  ultrasound measures of the bilateral Internal jugular vein with numeric blood flow characterization
Bilateral Internal jugular vein pressure | 2-3 hours
  ultrasound measures of the bilateral Internal jugular vein using a pressure measurement device
Bilateral Internal jugular vein area | 2-3 hours
  ultrasound measures of the bilateral Internal jugular vein to measure vein area

CONTACTS AND LOCATIONS:
Overall Officials: Stuart M Lee, PhD, Principal Investigator — National Aeronautics and Space Administration (NASA)
Locations (1):
- NASA, Houston, Texas, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-05-31): https://cdn.clinicaltrials.gov/large-docs/38/NCT06500338/ICF_000.pdf